CLINICAL TRIAL: NCT05735756
Title: Effect of Citalopram on Chest Pain in Patients With Functional Chest Pain
Acronym: Ci-FCP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The clinical trial has ended prematurely due to low patient recruitment
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof.dr. A.J. (Arjan) Bredenoord, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL77673.018.21
Record Dates: First submitted 2022-01-26; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Functional Chest Pain
MeSH Terms: interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citalopram 20mg (Active Comparator)
  Interventions: Drug: Citalopram 20mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citalopram 20mg — Citalopram 20mg once a day for 12 weeks
  Arms: Citalopram 20mg
Drug: Placebo — Placebo once a day for 12 weeks
  Arms: Placebo

SUMMARY:
Non-cardiac chest pain (NCCP) in the absence of musculoskeletal abnormalities, major esophageal motor disorders, gastroesophageal reflux or eosinophilic esophagitis is called functional chest pain (FCP). Most likely multiple factors play a role, such as esophageal hypersensitivity and enhanced perception. Citalopram and other antidepressants are proven to be effective in the treatment of functional gastrointestinal disorders such as irritable bowel syndrome. With this trial the investigators want to assess the effect of citalopram on symptoms of chest pain in patients with functional chest pain.

DETAILED DESCRIPTION:
Chest pain can be divided in cardiac or non-cardiac chest pain (NCCP). To establish the diagnosis NCCP, acute coronary disease has to be ruled out first. NCCP can be caused by functional chest pain (FCP). NCCP in the absence of musculoskeletal abnormalities, major esophageal motor disorders, gastroesophageal reflux or eosinophilic esophagitis is called FCP. The pathophysiology is not fully understood. Most likely multiple factors play a role, such as esophageal hypersensitivity and enhanced perception. Citalopram and other antidepressants are proven to be effective in the treatment of functional gastrointestinal disorders such as irritable bowel syndrome. However, available data regarding low dose antidepressants in functional chest pain is inconclusive. Moreover, all current evidence concerning the effect of low dose antidepressants in patients with functional chest pain is extracted from trials that pooled patients with different functional esophageal disorders. With this trial the investigators want to assess the effect of citalopram on symptoms of chest pain in patients with functional chest pain.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Minimum age: 18 years
* Functional chest pain according to Rome IV criteria
* Ruled out cardiac origin of chest pain
* ECG with corrected QT interval (QTc) within the normal range (<450ms male, <460ms female)
* Symptoms of chest pain for at least 6 months
* Frequency of symptoms at least once a week
* Gastroduodenoscopy, high-resolution manometry and 24-hour pH-impedance monitoring need to have been performed recently.

Exclusion Criteria:

* Currently using antidepressants
* Contraindication for the use of SSRI
* Already tried antidepressants off-label to treat chest pain
* Known allergy to citalopram
* Severe and clinically unstable concomitant disease
* Pregnant, lactating or fertile women (without contraception)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Global assessment of patient reported change in chest pain after 6 weeks of treatment. | 6 weeks after start of the study
  Patients will be asked; "Compared to the start of the treatment, how would you rate the chest pain now?
  * Completely resolved
  * Moderately better
  * Slightly better
  * No change
  * Slightly worse
  * Moderately worse
  * Much worse Patients who answered completely resolved or moderately better will be defined as treatment success.

SECONDARY OUTCOMES:
Global assessment of patient reported change in chest pain after 12 weeks of treatment. | 12 weeks after start of the study
  Patients will be asked; "Compared to the start of the treatment, how would you rate the chest pain now?
  * Completely resolved
  * Moderately better
  * Slightly better
  * No change
  * Slightly worse
  * Moderately worse
  * Much worse Patients who answered completely resolved or moderately better will be defined as treatment success.
Symptom frequency | Daily diary during the entire duration of the study (12 weeks)
  Patients are asked to report the frequency of symptom episodes on a daily base
Symptom severity | Daily diary during the entire duration of the study (12 weeks)
  Patients are asked to report the severity of every symptom episode on a daily base.
  The severity will be rated on a 4-point scale: mild (1, the symptom was well tolerated and did not last long) moderate (2, the symptom caused some discomfort, but did not interfere with usual activities), severe (3, the symptom caused a great deal of discomfort, and interfered with usual activities), disabling (4, the symptom was unbearable and interfered considerably with usual activities).
Chest pain will be scored on a 0-10 visual analog scale (VAS-score) | Baseline, 6 weeks and 12 weeks
  Patients are asked to report the severity of the chest pain every 6 weeks
Health related quality of life measured using 36-Item Short Form Health Survey (SF36) | Baseline, 6 weeks and 12 weeks
  The health related quality of life is measured every 6 weeks
Psychological comorbidity using the Hospital Anxiety and Depression Scale (HADS) | Baseline, 6 weeks and 12 weeks
  Psychological comorbidity is assessed every 6 weeks
Adverse events/side effects | Adverse event reporting period is defined as the period following time of written informed consent up to 3 months after end of the observation period.
  Patients are asked to report adverse events and side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No